CLINICAL TRIAL: NCT02450266
Title: Prospective Multicenter, Randomized Study Comparing the Diagnostic Efficacy of a Targeted MRI/Ultrasound Fusion-guided Prostate Biopsy Versus a Systematic Transrectal Ultrasound-guided Biopsy in Men With at Least on Negative Prostate Biopsy
Brief Title: Study Comparing MRI/Ultrasound Fusion-guided Prostate Biopsy Versus Systematic Transrectal Ultrasound-guided Biopsy
Acronym: PROFUSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: German Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 004
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Prostate Cancer
Keywords: Primary disease; multiparametric MRI; targeted prostate biopsy; MRI/ultrasound fusion-guided prostate biopsy; systematic transrectal ultrasound-guided prostate biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: Transrectal ultrasound-guided biopsy (Active Comparator): Patients of arm A receive a systematic transrectal ultrasound-guided prostate biopsy (12-18 biopsy cores depending on individual prostate volume)
  Interventions: Device: Systematic transrectal ultrasound-guided prostate biopsy
- B: MRI/ultrasound fusion-guided biopsy (Experimental): Patients of arm B receive a targeted MRI/ultrasound fusion-guided prostate biopsy. From each prostate lesion defined in the diagnostic multiparametric MRI two targeted biopsy cores will be taken.
  Interventions: Device: MRI/ultrasound fusion-guided prostate biopsy

INTERVENTIONS:
Device: Systematic transrectal ultrasound-guided prostate biopsy — 12-18 systematic biopsy cores
  Arms: A: Transrectal ultrasound-guided biopsy
Device: MRI/ultrasound fusion-guided prostate biopsy — 2 targeted biopsy cores from each prostate lesion
  Arms: B: MRI/ultrasound fusion-guided biopsy

SUMMARY:
Patients will be submitted to a multiparametric MRI examination of the prostate. Subsequently, all participants will be randomized (1:1) into both study arms. In study arm A patients will be submitted to the gold-standard which comprises systematic transrectal ultrasound-guided prostate biopsy. In study arm B patients will be submitted to targeted prostate biopsy based on the multiparametric MRI findings.

DETAILED DESCRIPTION:
In men with previously negative prostate biopsy and persistent elevated prostate-specific antigen (PSA) value, it is unclear which biopsy strategy offers the highest detection rate for significant prostate cancer. The hypothesis of this study is that targeted MRI/ultrasound fusion-guided biopsy improves the detection rates of significant prostate cancers compared with systematic transrectal ultrasound-guided prostate biopsy.

Men with at least one previously negative transrectal ultrasound-guided biopsy and persistently elevated PSA values (> 3 ng/ml) or PSA velocity >0.75 ng/ml/p.a. will be submitted to a multiparametric MRI examination of the prostate. Subsequently, all participants will be randomized (1:1) into both study arms. In study arm A patients will be submitted to the gold-standard which comprises systematic transrectal ultrasound--guided prostate biopsy. In study arm B patients will be submitted to targeted prostate biopsy based on the multiparametric MRI findings. Targeted biopsies will be performed using MRI/ultrasound fusion-guided.

ELIGIBILITY:
Inclusion Criteria:

* At least one negative transrectal ultrasound-guided prostate biopsy
* PSA > 3.0 ng/ml or PSA velocity >0.75 ng/ml/p.a.

Exclusion Criteria:

* Known prostate cancer
* PSA >50 ng/ml
* Previous MRI-targeted prostate biopsy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 586 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Detection rate of significant prostate cancers | One week after biopsy

SECONDARY OUTCOMES:
Overall detection rate of prostate cancers | One week after biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Christian Arsov, MD, Principal Investigator — Department of Urology, University Hospital Düsseldorf
Locations (3):
- Germany (3):
  - Department of Urology, Charité-Universitätsmedizin, Berlin
  - Department of Urology, University Hospital Düsseldorf, Düsseldorf
  - Department of Urology, University Hospital Jena, Jena